CLINICAL TRIAL: NCT01105169
Title: Personalized Prevention of Colorectal Cancer Trial (PPCCT)
Brief Title: Precision-Based Magnesium Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Qi Dai, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 100106
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
Keywords: Personalized prevention; Colorectal cancer; Investigational Nutrigenetic Studies; Magnesium; Gene polymorphism
MeSH Terms: conditions — Colorectal Neoplasms | interventions — magnesium diglycinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- GG genotype and magnesium treatment (Active Comparator): Participants who have the GG genotype will be assigned to magnesium glycinate.
  Interventions: Dietary Supplement: Magnesium glycinate
- GG genotype and placebo (Placebo Comparator): Participants who have the GG genotype will be assigned to placebo group
  Interventions: Dietary Supplement: Placebo
- GA/AA genotype and magnesium treatment (Active Comparator): Participants who have the GA/AA genotype will be assigned to magnesium glycinate
  Interventions: Dietary Supplement: Magnesium glycinate
- GA/AA genotype and Placebo (Placebo Comparator): Participants who have the GA/AA genotype will be assigned to placebo group
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium glycinate — Oral administration of magnesium glycinate daily for 12 weeks
  Arms: GA/AA genotype and magnesium treatment; GG genotype and magnesium treatment
Dietary Supplement: Placebo — Oral administration of identical-appearing placebo daily for 12 weeks
  Arms: GA/AA genotype and Placebo; GG genotype and placebo

SUMMARY:
Colorectal cancer is the fourth most common incident cancer and the second most common cause of cancer death in the United States, with approximately 150,000 new cases and 57,000 deaths per year. High calcium intake and magnesium may protect against colorectal cancer and adenoma, however, results have been inconsistent. We found that genetic makeup, associated with magnesium absorption and re-absorption, significantly interacted with the calcium and magnesium ratio in relation to the both adenomatous and hyperplastic polyps. Participants who carried at least one 1482Ile allele (G->A)of TRPM7 and who consumed diets with a high calcium/magnesium ratio were at a higher risk of adenoma and hyperplastic polyps than were participants who did not carry the polymorphism. We hypothesize that the reduction in the dietary Ca/Mg ratio may change the markers directly related to tumorigenesis. The primary aims of this study are to conduct a randomized placebo-controlled intervention trial to test whether reducing the Ca/mg intake ratio through magnesium supplementation has effects on the related biomarkers. We will also examine whether the effect of modulating Ca/Mg intake ratio may be more pronounced among those who carry the 1482Ile allele compared those who don't carry the 1482Ile allele. Results from our study will help to identify people at a high risk of colorectal adenoma and to develop personalized strategies to prevent occurrence of colorectal adenoma, and thus, colorectal cancer through dietary change or nutritional fortification.

ELIGIBILITY:
Inclusion Criteria:

* Hyperplastic polyp or/and Adenoma cases
* Polyps free participants with any of the following high risk of colorectal polyps or cancer: (1) family history of colorectal cancer or polyps; (2) current cigarette smoker; (3) obesity (BMI≥30 kg/m2); (4) low intake of fiber (lowest fiber intake quartile: daily intake <16.6g); (5) high intake of red meat and well-done or processed meat (mutageneity index ≥5852).
* Participants from the TCPS (IRB # 090235), the TIARS (IRB # 090235), from Vanderbilt University Hospital or from other resources
* Consent to be contacted for future studies in TCPS (IRB # 020462), TIARS (IRB#090235)
* Participants with a calcium intake ≥ 700 mg/day measuring with 24 hour dietary recalls
* Participants with a calcium intake < 2000 mg/day measuring with 24 hour dietary recalls
* Participants with a calcium/magnesium intake ratio > 2.6
* Participants with known genotype for Thr1482Ile polymorphism in TRPM7
* Will live in Nashville or surrounding area in the next 6 months

Exclusion Criteria:

* Intolerance to magnesium glycinate or microcrystalline cellulose (placebo)
* Chronic renal diseases and hepatic cirrhosis
* Chronic ischemic heart disease with unstable angina, chronic heart failure at class III or IV and acute myocardial infarction in the last 6 months
* Chronic diarrhea
* Current breastfeeding
* Current or planned pregnancy
* Type I diabetes mellitus
* Pituitary dwarfism
* Use of digoxin and licorice
* Current use of blood anticoagulant drugs such as Dicumarol(Warfarin), Clopidogrel (Plavix), Prasugrel HCl (Efficent), Ticlopidine (Ticlid), Lovenox (Enoxaparin), Fragmin (Dalteparin), Innohep (Tinzaparin), Eptifibatide (Integrilin), Tyrofiban (Aggrastat), and Abciximab (Reopro)
* Current use of lithium carbonate therapy (Eskalith, Lithobid, Lithonate, Lithotabs, Apo-Lithium carbonate, Apo-Lithium carbonate SR, Carbolth, Duralith, PMS-Lithium carbonate, PMS-Lithium citrate)
* Individuals with a history of colon resection or colectomy due to any reason
* Individuals with any history of cancer other than non-melanoma skin cancer
* Individual with history of any organ transplantation
* Individual with a history of gastric bypass due to any reason
* Individuals with Inflammatory bowel disease
* Individuals if creatinine clearance is < 50
* Currently institutionalized
* Homeless individual (address, telephone etc.)
* Unable to provide informed consent
* Any condition that in the opinion of the investigator raises concerns about protocol compliance

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2011-03-11 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
The protein expression levels of TRPM7, MLKL in colorectal mucosa | 12 week (rectal biopsies will be collected at the baseline and the end of the intervention)
  TRPM7 and MLKL have been detected using immunohistochemical (IHC) techniques.
Ratios of Ki67:BAX, Ki67:TUNEL (proliferation index) in rectal epithelial | 12 week (rectal biopsies will be collected at the baseline and the end of the intervention)
  Ki67:BAX and Ki67:TUNEL have been analyzed using immunohistochemical (IHC) techniques.
The expression of COX2 (inflammation) in rectal epithelia | 12 week (rectal biopsies will be collected at the baseline and the end of the intervention)
  COX2 has been analyzed using immunohistochemical (IHC)
The expression levels of apoptosis biomarkers (TUNEL and BAX) in colorectal mucosa | 12 week (rectal biopsies will be collected at the baseline and the end of the intervention)
  TUNEL and BAX were analyzed using immunohistochemical (IHC)

SECONDARY OUTCOMES:
Serum magnesium | 12 week
  Serum magnesium concentration was determined using 7D70 Magnesium Reagent Kit from Abbot Laboratories (Abbott Park, IL) the assay was conducted at the Vanderbilt Pathology Laboratory Services.
Post treatment body magnesium status | 12 week after treatment
  Body magnesium status obtained using magnesium tolerance test (MTT)
Circulation 25-Hydroxyvitamin D | 12 week
Serum C-reactive protein concentration | 12 week
  Assays of CRP for 180 participants were performed using immuno turbidimetric immunoassay based commercial assay kits (Pointe Scientific, Inc, Canton, MI) at Vanderbilt Lipid Laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Qi Dai, MD, PhD, Principal Investigator — Vanderbilt University Medical Center; Chang Yu, PhD, Principal Investigator — Vanderbilt University Medical Center; Martha J Shrubsole, Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Sun E, Zhu X, Ness RM, Murff HJ, Sun S, Yu C, Fan L, Azcarate-Peril MA, Shrubsole MJ, Dai Q. Magnesium treatment increases gut microbiome synthesizing vitamin D and inhibiting colorectal cancer: results from a double-blind precision-based randomized placebo-controlled trial. Am J Clin Nutr. 2025 Nov;122(5):1185-1194. doi: 10.1016/j.ajcnut.2025.09.011. Epub 2025 Sep 12. PMID 40946805
- [Derived] Sun S, Zhu X, Huang X, Yu C, Su T, Murff HJ, Ness RM, Azcarate-Peril MA, Shrubsole MJ, Dai Q. The Association of Gut Microbiota With TRPM7 Genotype, Colorectal Polyps, and Magnesium. J Nutr. 2025 Nov;155(11):3713-3725. doi: 10.1016/j.tjnut.2025.07.015. Epub 2025 Jul 30. PMID 40750038
- [Derived] Fan L, Zhu X, Sun S, Yu C, Huang X, Ness R, Dugan LL, Shu L, Seidner DL, Murff HJ, Fodor AA, Azcarate-Peril MA, Shrubsole MJ, Dai Q. Ca:Mg ratio, medium-chain fatty acids, and the gut microbiome. Clin Nutr. 2022 Nov;41(11):2490-2499. doi: 10.1016/j.clnu.2022.08.031. Epub 2022 Sep 12. PMID 36223712
- [Derived] Fan L, Zhu X, Rosanoff A, Costello RB, Yu C, Ness R, Seidner DL, Murff HJ, Roumie CL, Shrubsole MJ, Dai Q. Magnesium Depletion Score (MDS) Predicts Risk of Systemic Inflammation and Cardiovascular Mortality among US Adults. J Nutr. 2021 Aug 7;151(8):2226-2235. doi: 10.1093/jn/nxab138. PMID 34038556
- [Derived] Fan L, Yu D, Zhu X, Huang X, Murff HJ, Azcarate-Peril MA, Shrubsole MJ, Dai Q. Magnesium and imidazole propionate. Clin Nutr ESPEN. 2021 Feb;41:436-438. doi: 10.1016/j.clnesp.2020.12.011. Epub 2021 Jan 7. PMID 33487303